CLINICAL TRIAL: NCT03414411
Title: Addressing Alcohol/HIV Consequences in Substance Dependence - Boston ARCH Cohort: The 4F Study
Brief Title: Boston Alcohol Research Collaboration on HIV/AIDS (ARCH) Cohort: The 4F Study
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-35443; U01AA020784 (NIH)
Record Dates: First submitted 2017-10-30; First posted 2018-01-30 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: HIV Infections; Alcohol Drinking; Substance-Related Disorders; Bone Diseases; Falls Injury; Fractures, Bone; Injuries
Keywords: HIV; Alcohol Use; Substance Use; Bone Disease; Falls; Fractures
MeSH Terms: conditions — HIV Infections; Alcohol Drinking; Substance-Related Disorders; Bone Diseases; Fractures, Bone; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — saliva
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to follow a cohort of HIV-infected adults who have alcohol and/or drug use to: 1) test the associations between alcohol (and illicit drugs and polypharmacy (multiple prescribed medications)) and falls (fractures secondarily), and whether frailty mediates these associations; and 2) test the associations between alcohol (and illicit drugs and polypharmacy) and utilization (emergency department use and hospitalization for falls and fractures), and whether frailty mediates them.

To achieve the stated aims the investigators will expand (to 400) and continue to follow an existing prospective cohort (The Boston ARCH Cohort) of adults with HIV infection and a high prevalence of exposure to alcohol, other drugs, and polypharmacy. The Boston ARCH Cohort is a longitudinal cohort (1-3.5 years of follow-up) of 250 HIV-infected men and women with current substance dependence or ever injection drug use that have a spectrum of alcohol use.

DETAILED DESCRIPTION:
Up to a third of middle-aged people living with HIV infection (PLWH) experience falls each year. Falls are the most common cause of non-fatal injury in the US and the cost from emergency department visits and hospitalizations are enormous. PLWH are more susceptible to falls and their serious consequences because 1) despite control of HIV viremia, inflammation persists and underlies HIV-associated comorbidities and complications that occur at a relatively young age (so-called premature aging); 2) specific comorbidities (e.g., neuropathy, osteoporosis) and complications (e.g., frailty and impaired physical function) make falls more likely and recovery from them more difficult; 3) alcohol use exacerbates inflammation, and may increase risk for comorbidities and complications; and 4) alcohol use, illicit drug use and polypharmacy can increase the likelihood of a fall. Despite this, fall prevention has not been extensively studied among PLWH. Interventions are needed to address falls in PLWH but none have been tailored for this population. Understanding risk factors and targets for intervention among PLWH are essential; cohort studies can provide the information needed for intervention development.

This study is part the Consortia for HIV/AIDS and Alcohol-Related Research Trials (CHAART). It describes the continuation and expansion of a cohort that is one of three in the Uganda Russia Boston Alcohol Network for Alcohol Research Collaboration on HIV/AIDS (URBAN ARCH). The URBAN ARCH theme is to address consequences of alcohol use on HIV-associated comorbidities and complications to increase treatment availability and improve outcomes. In line with that theme the investigators will continue to follow and expand (to 400) an existing cohort of PLWH and a high prevalence of exposure to alcohol, illicit drugs, and polypharmacy (the Boston ARCH Cohort) in the Frailty, Functional impairment, Falls, and Fractures (4F study) to: (in 2 Primary Aims) 1) Test the associations between alcohol (and illicit drugs and polypharmacy) and falls (fractures secondarily); and 2) Test the associations between alcohol (and illicit drugs and polypharmacy) and acute healthcare utilization (emergency department use and hospitalization for falls and fractures). The investigators will examine the role frailty plays in these associations between alcohol, drugs and medications and the aforementioned clinical and utilization outcomes. By achieving these aims the investigators will gain substantially greater understanding of these comorbidities and complications in PLWH exposed to alcohol and other psychoactive substances; this knowledge will serve to inform the development of ways to identify, prevent and manage falls, fractures, frailty and functional impairment.

ELIGIBILITY:
Inclusion Criteria:

* Ability to speak English (fluency)
* Willing to provide information for >1 contact person likely to know their whereabouts for follow-up.
* Documented HIV antibody by ELISA confirmed by Western Blot or current HIV viral load greater than 10,000 (in any medical record); or HIV antibody by 4th generation ELISA confirmed by a "Multi-Spot" rapid test for discrimination of HIV-1 from HIV-2 infection and, if necessary in the case of discordant results, nucleic acid testing (NAT) for HIV-1; or any other confirmatory pathway approved by the Massachusetts Department of Public Health, U.S. Centers for Disease Control and Prevention or BMC Center for Infectious Diseases.
* Any past 12 month use of illicit drugs, marijuana (not recommended by a healthcare provider), or nonmedical use of prescription medications (assessed using the Tobacco, Alcohol, Prescription Medication and Other Substances (TAPS) Tool); OR past 12 month alcohol use with positive AUDIT-C score (≥3 for females and ≥4 for males)
* OR, an existing participant in the Boston ARCH Cohort

Exclusion Criteria:

* Inability to consent or understand interview (determined by trained research assistant)
* Under age 18
* Plans to leave Boston area in <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All existing Boston ARCH Cohort participants will be offered enrollment into the 4F Study, a continuation of the Boston ARCH Cohort; additional participants will be identified from adult primary care and HIV clinics Boston Medical Center and Boston Healthcare for the Homeless Program (BHCHP).
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2022-11-09 (Actual); Study Completion 2023-04-27 (Actual)

PRIMARY OUTCOMES:
Any self-reported falls | 6-month window prior to study entry and 6-month window prior to each annual visit, for up to 3.5 years
  The primary outcome for Aim 1 analyses is any self-reported falls, with falls defined as an unexpected event, including a slip or trip, in which a participant lost their balance and landed on the floor, ground, or lower level, or hit an object such as a table or chair.
Healthcare utilization | 6-month window prior to study entry and 6-month window prior to each annual visit, for up to 3.5 years
  We will use self-report to measure recent emergency department use and hospitalization for falls and fractures.

SECONDARY OUTCOMES:
Falls from electronic medical record review [Time Frame: 6 months prior to study entry and prior to each annual visit] Electronic records will identify falls that receive medical attention. Falls from electronic record review | 6-month window prior to study entry and 6-month window prior to each annual visit, for up to 3.5 years
  Electronic records will identify falls that receive medical attention.
Self-reported fractures | 6-month window prior to study entry and 6-month window prior to each annual visit, for up to 3.5 years
  Fractures, while less common than falls, are significant events that will be assessed primarily through self-report.
Fractures from electronic medical record review | 6-month window prior to study entry and 6-month window prior to each annual visit, for up to 3.5 years
  Electronic record review, including attention to a subset associated with fragility, will identify self-reported fractures.
Healthcare utilization | 12-month window prior to study entry and 12-month window prior to each annual visit, for up to 3 years
  Self-reported hospitalizations and emergency department visits will be identified using electronic medical records.

OTHER OUTCOMES:
Frailty | Between study entry and final visit, measured annually, for up to 3 years
  The frailty phenotype includes measures of exhaustion, low activity, weight loss, slowed walking, weak grip.
Impaired physical function | Between study entry and final visit, measured annually, for up to 3 years
  Balance, gait, strength and endurance in standing, walking, and chair rise tests, will be measured using the Short Physical Performance Battery.

CONTACTS AND LOCATIONS:
Overall Officials: Theresa W Kim, MD, Principal Investigator — Boston University
Locations (1):
- Boston University Medical Campus, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided